CLINICAL TRIAL: NCT03400969
Title: A Randomized Controlled Trial of the Effectiveness of Three Different Oral Moisturizers in Palliative Care Patients.
Brief Title: Effectiveness of Three Different Oral Moisturizers in Palliative Care Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2016/2316
Record Dates: First submitted 2017-12-14; First posted 2018-01-17 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-01

CONDITIONS: Xerostomia
Keywords: Palliative; Moisturisers; Dry mouth; Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: The different moisturizers will be compared in a double blind, cross-over design. Patient responses will be collected at baseline, immediately after exposure and after 2 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Block randomisation is made by a person, other than the one who applies the product. Neither the patient nor the person who records the product or the person who registers data knows which product is used for the intervention. The product is not labeled with name
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glycerol 17 % (Active Comparator): Oral moisturizer
  Interventions: Device: Glycerol 17%
- Aequasyal (OGT) (Active Comparator): Oral moisturizer
  Interventions: Device: Aequasyal (OGT)
- Salient (new product) (Active Comparator): Oral moisturizer
  Interventions: Device: Salient (new product)

INTERVENTIONS:
Device: Glycerol 17% — Glycerol will be applied, using gauze on a lockable tweezer, at the end of the oral care procedure performed by a dentist.
  Arms: Glycerol 17 %
Device: Aequasyal (OGT) — Aequasyl (OGT) will be sprayed on the mucosa, at the end of the oral care procedure, preformed by a dentist.
  Arms: Aequasyal (OGT)
Device: Salient (new product) — Salient (new Product) will be applied/given on a spoon, at the end of the oral care procedure, preformed by a dentist.
  Arms: Salient (new product)

SUMMARY:
This study compares the effectiveness of 3 different oral moisturizers; 17% watery solution of glycerol, OGT oral spray, Aequasyal, and a newly developed Product, Salient.

DETAILED DESCRIPTION:
Background:

A majority of patients in palliative care have problems with dry mouth caused by medication or as a direct result of the mortal condition. Dry mouth will cause a variety of problems that commonly affect the disease negatively and contribute to reduced quality of life in the patient's last stage of life. A Cochrane review from 2011 concludes that "there are several moisturising agents available, but no strong evidence that any topical therapy is effective for relieving the symptom of dry mouth." It also concludes that "Oxygenated glycerol triester (OGT) oral spray is more effective than an aqueous electrolyte spray."1

Objectives:

To compare the effectiveness of 3 different oral moisturisers, ; 17 % watery solution of glycerol, OGT oral spray, Aequasyal® and a newly developed product, Salient®.

Methods/design:

30 patients will be recruited from a Norwegian palliative care unit. Eligibility criteria for participants are:

1. The patients have xerostomia (subjective feeling of dry mouth). 2
2. The patients are palliative and in institutionalized care.
3. Curative treatment of existing diseases has been completed.
4. WHOs functional status 3/Karnofsky functional status 30 - 40 % (only capable of limited self-care, tied to bed or chair more than 50% of wake time).3, 4
5. Participants are cognitively functioning, capable of and willing to consent, capable of giving responses to a limited questionnaire and are expected to remain at the care centre for a minimum of 3 days.

Patients treated with radiotherapy in head and neck region, are excluded from this trial.

The different moisturizers will be compared in a double blind, cross-over design. All patients will be randomized to all three treatments in the cross-over trial, with a minimum of 24 hours wash-out period between the treatments. Patient responses will be collected at baseline, immediately after exposure and after 2 hours. Medical history and medication will be recorded. Primary outcome variables are the subjective feeling of xerostomia, pain/discomfort and speech disturbance.

Ethical considerations:

An application for approval of this study will be sent to the Regional Ethical Committee (REC). There are no known side effects of the agents or methods that will be applied.

Discussion:

To the investigators knowledge, the proposed randomized controlled trial of the effect of three different oral moisturizers will be the first study of this kind to be performed in patients in palliative institutionalized ward. There are no known adverse effects of the products used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The patients have xerostomia (subjective feeling of dry mouth). 2
2. The patients are palliative and in institutionalized care.
3. Curative treatment of existing diseases has been completed.
4. WHOs functional status 3/Karnofsky functional status 30 - 40 % (only capable of limited self-care, tied to bed or chair more than 50% of wake time).
5. Participants are cognitively functioning, capable of and willing to consent, capable of giving responses to a limited questionnaire and are expected to remain at the care centre for a minimum of 3 days.

Exclusion Criteria:

Patients treated with radiotherapy in head and neck region.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Subjective xerostomia | 3 days
  Measured on a 5-point Likert-scale:
  Subjective feeling of dry mouth:
  1. Not dry
  2. Insignificantly dry
  3. Fairly dry
  4. Almost completely dry
  5. Completely dry

SECONDARY OUTCOMES:
Pain/discomfort | 3 days
  Measured on a 5-point Likert-scale:
  Subjective feeling pain/discomfort:
  1. No pain
  2. Insignificant pain/discomfort
  3. Some pain/discomfort
  4. Much pain/discomfort
  5. Strong pain/discomfort
Speech | 3 days
  Measured on a 5-point Likert-scale:
  Xerostomia regarding impact on ability to speak:
  1. Not difficulties
  2. Insignificant difficulties
  3. Some difficulties
  4. Significant difficulties
  5. Major difficulties
Diurnal variation | 3 days
  Measured on a 5-point Likert-scale:
  At what times are xerostomia most pronounced:
  1. At night
  2. In the morning
  3. In the afternoon
  4. In the evening
  5. No diurnal difference
Situational dry mouth | 3 days
  Measured on a 3-point Likert-scale:
  1. By intake of medication
  2. By worsening of the disease
  3. In Connection with thirst

CONTACTS AND LOCATIONS:
Overall Officials: Gunhild V Strand, DDS, PhD, Principal Investigator — University of Bergen, Norway
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be available by request after publication of effect article.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after publication of article.